CLINICAL TRIAL: NCT00476359
Title: Lopinavir/r Plus Saquinavir Salvage Therapy in HIV-infected Children With NRTI and/or NNRTI Failure: PK and Two-year Treatment Follow up
Brief Title: A PK and Salvage Study for Children With HIV-infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Roche for trial and Saquinavir,and Abbott for Kaletra (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 017
Record Dates: First submitted 2007-05-20; First posted 2007-05-22 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infections
Keywords: Lopinavir/r; Saquinavir; Dual boosted PIs; Pharmacokinetics; HIV children; C min; Second line HAART; ARV; VL failure; Dosage; To evaluate treatment response; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Saquinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- double-boosted PI (Other): double-boosted protease inhibitor combination
  Interventions: Drug: Lopinavir/r plus saquinavir

INTERVENTIONS:
Drug: Lopinavir/r plus saquinavir — lopinavir/ritonavir 230/57.5 mg/m2 orally twice daily and saquinavir 50 mg/kg orally twice daily

SUMMARY:
To evaluate the pharmacokinetics (PK) of LPV/r with saquinavir in HIV-1 infected children. To evaluate treatment response (clinical, immunological and virological) to LPV/r, SQV in Thai children.

DETAILED DESCRIPTION:
The PK and 24 week data has been published in Pediatric Infectious Diseases Journal. It showed that plasma drug concentrations of saquinavir, lopinavir and ritonavir were at the higher limits of expected ranges for adult treatment at approved dosages (1000/100 mg BID for saquinavir, 400/100 mg BID for lopinavir/r). The regimen was well tolerated and showed significant CD4 rise and VL decline at 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV-1 infection by HIV-DNA PCR if < 18 months old or by HIV ELISA if greater than or equal to 18 months old
2. Subject is less than or equal to 16 years of age at the day of the first dosing.
3. Subject is failing a current NRTI and/or NNRTI containing regimen and is naïve to protease inhibitor containing therapy.
4. Results of biochemistry and haematology testing should be within pre-specified ranges.
5. Subject is able to swallow capsules
6. Caretaker(s) is/are able and willing to sign the Informed Consent Form prior to screening evaluations.

Exclusion Criteria:

1. History of sensitivity/idiosyncrasy to lopinavir, ritonavir, saquinavir or chemically related compounds or excipients which may be employed in the trial.
2. Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
3. Inability of both child and caregiver(s) to understand the nature and extent of the trial and the procedures required.
4. Use of any of concomitant medication, including the drug listed below, that may interfere with the pharmacokinetics of LPV/r or SQV.

   * NNRTIs
   * Rifampicin
   * Rifabutin
   * Phenobarbital
   * Phenytoine
   * Carbamazepine
   * Dexamethasone
   * Ketoconazole
   * Clarithromycin
5. Pregnancy

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2003-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Intensive 0-12h PK sampling for plasma levels of LPV and SQV, and blood sampling. CD4 viral load safety lab every 3 months. | 96 week

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — HIV-NAT, Bangkok, Thailand; Pope Kosalaraksa, MD, Principal Investigator — Khon Kaen University
Locations (3):
- Thailand (3):
  - Chulalongkorn University Hospital, Department of Pediatrics, Bangkok, Bangkok
  - The HIV Netherlands Australia Thailand Research Collaboration, Bangkok, Bangkok
  - Khon Kaen University, Khon Kaen, Changwat Khon Kaen

REFERENCES:
- [Result] Ananworanich J, Kosalaraksa P, Hill A, Siangphoe U, Bergshoeff A, Pancharoen C, Engchanil C, Ruxrungtham K, Burger D; HIV-NAT 017 Study Team. Pharmacokinetics and 24-week efficacy/safety of dual boosted saquinavir/lopinavir/ritonavir in nucleoside-pretreated children. Pediatr Infect Dis J. 2005 Oct;24(10):874-9. doi: 10.1097/01.inf.0000180578.38584.da. PMID 16220084
- [Result] Kosalaraksa P, Engchanil C, Bunupuradah T, Luesomboon W, Sunthornkachit R, Bunruen S, Intasan J, Jupimai T, Hirunwadee N, Lumbiganon P, Ruxrungtham K on behalf of the PREDICT study team. Prevalence of anemia and impact of iron status in Thai and Cambodian HIV infected children with moderate immunosuppression (PREDICT study), poster No. TUPEB 137. Poster presented at the 4th International AIDS Society Conference on HIV Pathogenesis, Treatment and Prevention, Sydney, Australia, July 22-25, 2007
- [Result] Jasper van der Lugt, Torsak Bunupuradah, Pope Kosalaraksa, Thanyawee Puthanakit, Chulapan Engchanil, Waraporn Sakornjun, Meena Gorowara, ROCHE, Kiat Ruxrungtham, David Burger, Jintanat Ananworanich: Therapeutic Drug Monitoring of lopinavir and saquinavir in Thai HIV infected Children. Poster will be presented at the 15th Conference on Retroviruses and Opportunistic Infections, Boston, USA, February 3-7, 2008.
- [Result] Torsak Bunupuradah, Pope Kosalaraksa, Chulapan Engchanil, Pitch Boonrak, Tawan Hirunyanulux, Sasiwimol Ubolyam, Pagakrong Lumbiganon, Kiat Ruxrungtham, Emily Labriola-Tompkins, Jintanat Ananworanich, and HIV-NAT 017 Study Team: Efficacy and safety of double boosted SQV/LPV/r combination at 96 weeks in Thai children who have failed NRTI/NNRTI-.based regimens. Abstract # R-143. Abstract will be presented at the 15th Conference on Retroviruses and Opportunistic Infections, Boston, USA, February 3-7, 2008.
- [Result] Bunupuradah T, van der Lugt J, Kosalaraksa P, Engchanil C, Boonrak P, Puthanakit T, Mengthaisong T, Mahanontharit A, Lumbiganon P, Tompkins E, Burger D, Ruxrungtham K, Ananworanich J; HIV-NAT 017 Study Team. Safety and efficacy of a double-boosted protease inhibitor combination, saquinavir and lopinavir/ritonavir, in pretreated children at 96 weeks. Antivir Ther. 2009;14(2):241-8. PMID 19430099
- [Result] Kosalaraksa P, Bunupuradah T, Engchanil C, Boonrak P, Intasan J, Lumbiganon P, Burger D, Ruxrungtham K, Schutz M, Ananworanich J; HIV-NAT 017 Study Team. Double boosted protease inhibitors, saquinavir, and lopinavir/ritonavir, in nucleoside pretreated children at 48 weeks. Pediatr Infect Dis J. 2008 Jul;27(7):623-8. doi: 10.1097/INF.0b013e31816b4539. PMID 18520443
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org